CLINICAL TRIAL: NCT02671903
Title: AV Optimisation Delivered With Direct His Bundle Pacing, in Patients With Heart Failure, Long PR Without Left Bundle Branch Block: Randomised Multi-centre Clinical Outcome Study.
Brief Title: The His Optimised Pacing Evaluated for Heart Failure Trial (HOPE-HF).
Acronym: HOPE-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: British Heart Foundation (Other); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 15HH2828
Record Dates: First submitted 2016-01-26; First posted 2016-02-02 (Estimated); Results first posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pacemaker: AV optimised, His pacing (Active Comparator): Subjects will remain in this arm for 6 months before being crossed-over. See below intervention details.
  Interventions: Device: Pacemaker: AV optimised, His pacing.
- No pacing (No Intervention): Subjects will remain in this arm for 6 months before being crossed-over. The pacemaker will be programmed to VVI 30 bpm. Dynamic AV delay will be programmed off throughout the study.

INTERVENTIONS:
Device: Pacemaker: AV optimised, His pacing. — Direct His bundle pacing: a Medtronic Select Secure 3830 pacing lead will be positioned at the His bundle. If selective direct His bundle pacing cannot be achieved then non-selective His bundle pacing will be accepted. AV delay optimisation: will be performed using acute non-invasive blood pressure acquired using the Finometer device (Finapres Medical systems, Netherlands).
  Arms: Pacemaker: AV optimised, His pacing

SUMMARY:
This is a multi-centre, prospective randomised double-blinded cross over study, recruiting a sub-population of patients with heart failure.

All patients will be implanted with a CRT (Cardiac Resynchronisation Therapy) pacemaker with one of the leads positioned on the His bundle in order to obtain direct His-bundle capture. There will be a 2-month run-in period where the device is not active.

A double-blinded cross-over design will then be employed to investigate the effect of His bundle pacing. Patients will be allocated in random order to six month treatment periods in each of the following two states (1) No pacing; (2) AV optimised direct His-bundle pacing. Endpoint measurements will be taken at baseline, 6 months and 12 months post randomisation. Treatment allocation will be blinded to the endpoint assessor and the patient.

126 patients will be needed to detect the expected effect size on the primary endpoint with 90% power. A total of 160 patients will be recruited to allow for patient drop-out.

DETAILED DESCRIPTION:
Patients entering the study will attend for implantation of a CRT pacemaker device with one lead positioned on the His bundle. This will be performed either at the patient's local hospital or at Imperial College NHS healthcare Trust, no later than 4 months after the patient's screening visit.

All patients will be implanted with a Pacemaker or Implantable cardioverter defibrillator (ICD). In all patients a pacing lead will be positioned in the right atrium (typically the right atrial appendage). All patients will have a pacemaker lead positioned on the His bundle in order to obtain direct His-bundle capture. If it is not possible to successfully implant a His-bundle lead with selective direct His bundle capture or non-selective capture with < 40ms prolongation of the QRS duration, then a lead will be implanted in a lateral branch of the coronary sinus.

In patients who do not have an indication for an Implantable cardioverter defibrillator (ICD) a second ventricular lead will be implanted in a lateral branch of the coronary sinus. If direct His pacing has not been successfully achieved then a further lead will be positioned at the RV apex. In patients who do have an indication for an Implantable cardioverter defibrillator the ICD lead will be positioned in the right ventricle (either RV apex or RV septum).

AV delay optimisation will be performed using acute non-invasive blood pressure acquired using the Finometer device (Finapres Medical systems, Netherlands). The BHF (British Heart Foundation) alternation protocol will be used in order to minimise the effect of background noise.

After implantation of the device there will be a 2 month run-in period prior to randomisation, the device will be programmed not to deliver His bundle pacing therapy during this period.(Back up only pacing and defibrillator function will be enabled).

Two months after patients are implanted with their device, patients will be randomised to either receive active pacing treatment or back up only pacing (pacemaker programmed to VVI 30 bpm). After a further 6 months they will be crossed over to the alternative treatment arm. Treatment allocation will be obtained using an Interactive Web Response System (IWRS) programmed with a randomisation schedule provided by the trial statistician. Appropriate blocking will be used.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or above
* Ventricular Ejection Fraction (EF) < 40%; BNP needs to be ≥250ng/L for patients with EF 36-40%
* New York Heart Association (NYHA) class II-IV
* PR interval ≥200ms
* Narrow QRS duration (≤140ms) or prolonged QRS duration with typical Right Bundle Branch Block (RBBB) morphology on 12 lead ECG and sinus rhythm

Exclusion Criteria:

* Permanent or persistent atrial fibrillation (AF)
* Paroxysmal atrial fibrillation with history of sustained AF (more than 24 hours) in the 6 months prior to screening
* Patients who are unable to perform cardiopulmonary exercise testing
* Other serious medical condition with life expectancy of less than 1 year
* Lack of capacity to consent
* Pregnancy
* Contraindication to use of the relevant study device or leads (as per current manuals from manufacturer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Whinnett, BMBS MRCP, Principal Investigator — Senior Lecturer, Consultant Cardiologist and Electrophysiologist
Locations (15):
- United Kingdom (15):
  - West Hertfordshire Hospitals NHS Trust, Watford, Hertfordshire
  - Basildon and Thurrock Hospitals NHS Foundation Trust, Basildon
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Western Sussex Hospitals NHS Foundation Trust, Chichester
  - Medway NHS Foundation Trust, Gillingham
  - University Hospitals of Leicester NHS Trust, Leicester
  - Hammersmith Hospital, London
  - Barts Health NHS Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - Royal Brompton & Harefield NHS Foundation Trust, London
  - Papworth Hospital NHS Foundation Trust, Papworth Everard
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Great Western Hospitals NHS Foundation Trust, Swindon

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication. The data set will be created as an anonymised data sharing package and will be available post publication of data.
Supporting Information: Study Protocol, SAP
Time Frame: 6 months post publication of data
Access Criteria: The anonymised data set will be shared with the journal in which the papers are published.
  We will make the data available for analysis by non-commercial researchers on request to the Chief investigator.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients have a pacemaker device implanted and are subject to a 2-month run-in phase prior to randomisation.
Groups:
- Arm A: Pacing Followed by No-Pacing: Following a lead-in period of No-Pacing subjects will be placed under Direct His bundle pacing before being crossed-over to No-Pacing.
  See below intervention details.
  Pacing: AV optimised, His pacing.: Direct His bundle pacing: a Medtronic Select Secure 3830 pacing lead will be positioned at the His bundle. If selective direct His bundle pacing cannot be achieved then non-selective His bundle pacing will be accepted. AV delay optimisation: will be performed using acute non-invasive blood pressure acquired using the Finometer device (Finapres Medical systems, Netherlands).
  No-Pacing: The pacemaker will be programmed to VVI 30 bpm. Dynamic AV delay will be programmed off throughout the study.
- Arm B: No-Pacing Followed by Pacing: Following a lead-in period of No-Pacing subjects will be placed under No-Pacing before being crossed-over to Direct His bundle pacing.
  See below intervention details.
  No-Pacing: The pacemaker will be programmed to VVI 30 bpm. Dynamic AV delay will be programmed off throughout the study.
  Pacing: AV optimised, His pacing.: Direct His bundle pacing: a Medtronic Select Secure 3830 pacing lead will be positioned at the His bundle. If selective direct His bundle pacing cannot be achieved then non-selective His bundle pacing will be accepted. AV delay optimisation: will be performed using acute non-invasive blood pressure acquired using the Finometer device (Finapres Medical systems, Netherlands).
- Run-In Phase (Pre-Randomisation): 2-month run-in period for ALL patients post implantation of pacemaker. Set at No-Pacing.
Period: Period 0 (Run-In)
Arm/Group | Arm A: Pacing Followed by No-Pacing | Arm B: No-Pacing Followed by Pacing | Run-In Phase (Pre-Randomisation)
Started | 0 | 0 | 183 (Any patient that fails to the complete the run-in period are subsequently not randomised to a treatment Arm.)
Completed | 0 | 0 | 167
Not Completed | 0 | 0 | 16
Not completed — Death | 0 | 0 | 3
Not completed — Physician Decision | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 4
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Implantation Failure | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Period: Period 1 (Month 0 to Month 6)
Arm/Group | Arm A: Pacing Followed by No-Pacing | Arm B: No-Pacing Followed by Pacing | Run-In Phase (Pre-Randomisation)
Started | 83 (Post Randomisation, Patients now allocated to Arm A or Arm B) | 84 (Post Randomisation, Patients now allocated to Arm A or Arm B) | 0 (Post Randomisation, Patients now allocated to Arm A or Arm B)
Completed | 73 | 77 | 0 (Post Randomisation, Patients now allocated to Arm A or Arm B)
Not Completed | 10 | 7 | 0
Period: Period 2 (Month 6 to Month 12)
Arm/Group | Arm A: Pacing Followed by No-Pacing | Arm B: No-Pacing Followed by Pacing | Run-In Phase (Pre-Randomisation)
Started | 73 | 77 | 0 (Post Randomisation, Patients now allocated to Arm A or Arm B)
Completed | 67 | 69 | 0 (Post Randomisation, Patients now allocated to Arm A or Arm B)
Not Completed | 6 | 8 | 0

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Pacing Followed by No-Pacing | Arm B: No-Pacing Followed by Pacing | Total
Number analyzed (Participants) | 83 | 84 | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (9.03) | 68.0 (10.19) | 69.0 (9.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 74 | 77 | 151
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Asian | 10 | 7 | 17
  Ethnicity: Black | 3 | 5 | 8
  Ethnicity: Mixed | 0 | 2 | 2
  Ethnicity: Other Ethnic Group | 2 | 1 | 3
  Ethnicity: White | 68 | 69 | 137
Weight [Mean (Standard Deviation); unit: kg] | 85.22 (16.788) | 89.24 (17.636) | 87.24 (17.286)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.498 (5.0208) | 29.665 (5.5027) | 29.085 (5.2853)
Diastolic BP [Mean (Standard Deviation); unit: mmHg] | 69.0 (11.22) | 70.8 (11.31) | 69.9 (11.26)
Systolic BP [Mean (Standard Deviation); unit: mmHg] | 121.3 (19.07) | 121.7 (20.24) | 121.5 (19.61)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Exercise Capacity.
Description: Measured using peak oxygen uptake (VO2).
Time Frame: Baseline, 6 months and 12 months post randomisation.
Population: ITT
Measure: Mean (95% Confidence Interval); unit: ml/min/kg
Groups:
- Pacing: Pacing: AV optimised, His pacing.: Direct His bundle pacing: a Medtronic Select Secure 3830 pacing lead will be positioned at the His bundle. If selective direct His bundle pacing cannot be achieved then non-selective His bundle pacing will be accepted. AV delay optimisation: will be performed using acute non-invasive blood pressure acquired using the Finometer device (Finapres Medical systems, Netherlands).
- No-Pacing: No-Pacing: The pacemaker will be programmed to VVI 30 bpm. Dynamic AV delay will be programmed off throughout the study.
Arm/Group | Pacing | No-Pacing
Number analyzed (Participants) | 167 | 167
ml/min/kg | 14.0 [13.0 to 15.0] | 13.7 [12.8 to 14.6]
Statistical Analysis 1: Comparison: Pacing vs No-Pacing; Change in treatment effect taken from mixed-model output; Test type: Superiority; p = 0.3, Mixed Models Analysis; Fixed Effect for Treatment = 0.25, 95% CI 2-sided [-0.23 to 0.73]

2. Secondary Outcome: Changes in Echocardiographic Measurement of Left Ventricular Function (Ejection Fraction)
Description: Measured during echocardiogram.
Time Frame: Baseline, 6 months and 12 months post randomisation.
Population: ITT Population
Measure: Mean (95% Confidence Interval); unit: % (LVEF)
Arm/Group | Pacing | No-Pacing
Number analyzed (Participants) | 167 | 167
% (LVEF) | 33.4 [31.2 to 35.7] | 33.0 [31.0 to 34.9]

3. Secondary Outcome: Changes in B-type Naturietic Peptide (BNP).
Description: Measured from blood sample. Note: BNP was log-transformed before analysis in the mixed-model and then back transformed for presentation
Time Frame: Baseline, 6 months and 12 months post randomisation.
Population: ITT
Measure: Mean (95% Confidence Interval); unit: (ng/L)
Arm/Group | Pacing | No-Pacing
Number analyzed (Participants) | 167 | 167
(ng/L) | 323 [242 to 431] | 335 [257 to 436]

4. Secondary Outcome: Changes in Quality of Life Scores. - Minnesota
Description: Measured using Minnesota Score obtained from the Minnesota Living with Heart Failure Questionnaire (MLHFQ).
  Score range: 0 to 105, with higher scores indicating a worse outcome with more significant impairment in health-related quality of life
Time Frame: Baseline, 6 months and 12 months post randomisation.
Population: ITT - Note that some patients were not able to be analysed due to providing no questionnaire data.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Groups:
- No-Pacing: Following a lead-in period of No-Pacing subjects will be placed under No-Pacing before being crossed-over to Direct His bundle pacing
Arm/Group | Pacing | No-Pacing
Number analyzed (Participants) | 151 | 151
scores on a scale | 30.9 [25.1 to 36.7] | 34.6 [29.8 to 39.3]

5. Secondary Outcome: Cost Effectiveness Analysis (Using a Custom Designed Resource Utilisation Questionnaire)
Description: The analysis will be based on an intention-to-treat (ITT) principle. The economic evaluation will compare incremental costs and incremental outcomes of the direct His-bundle pacing against the standard medical care. The study will be performed from a societal perspective, which takes all relevant cost-categories and effects into account. The economic evaluation will consist of two parts, a cost-effectiveness analysis (CEA) and a cost utility analysis (CUA). In the CEA the incremental cost-effectiveness ratio (ICER) will be expressed as the incremental costs per point improvement in exercise capacity in peak VO2. The primary outcome measure in the CUA will be Qualitative Adjusted Life Years (QALYs), based on the EQ5D and Minnesota questionnaire scores.
  NOTE: Cost effectiveness was unable to be completed for HOPE-HF and as such null results are displayed
Time Frame: Baseline.
Population: NOTE: Cost effectiveness was unable to be completed for HOPE-HF and as such null results are displayed
Groups:
- ARM A (Pacemaker: AV Optimised, His Pacing --> No PAcing): Subjects will remain in this arm for 6 months before being crossed-over. See below intervention details.
  Pacemaker: AV optimised, His pacing.: Direct His bundle pacing: a Medtronic Select Secure 3830 pacing lead will be positioned at the His bundle. If selective direct His bundle pacing cannot be achieved then non-selective His bundle pacing will be accepted. AV delay optimisation: will be performed using acute non-invasive blood pressure acquired using the Finometer device (Finapres Medical systems, Netherlands).
- ARM B (No Pacing --> Pacemaker: AV Optimised, His Pacing): Subjects will remain in this arm for 6 months before being crossed-over. The pacemaker will be programmed to VVI 30 bpm. Dynamic AV delay will be programmed off throughout the study.
Arm/Group | ARM A (Pacemaker: AV Optimised, His Pacing --> No PAcing) | ARM B (No Pacing --> Pacemaker: AV Optimised, His Pacing)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Changes in Percentage Pacing
Description: Measured at completion of periods 1 & 2 (M6 & M12) - Percentage of time where device recorded ventricular pacing during each treatment period. Values are recorded across both arms.
  Results are descriptive and displayed by treatment and by period.
Time Frame: Baseline, 6 months and 12 months post randomisation.
Population: ITT - Note that results are presented per sequence (e.g, by arm per study period) due to the nature of this particular endpoint. Outcome is based on when participants are on Pacing therapy and as such a per-protocol analysis would read zero for any period when not on pacing.
Measure: Mean (Standard Deviation); unit: % (of time over period)
Groups:
- Arm A: Pacing Followed by No-Pacing: Following a lead-in period of No-Pacing subjects will be placed under Direct His bundle pacing before being crossed-over to No-Pacing.
  See below intervention details.
  Pacing: AV optimised, His pacing.: Direct His bundle pacing: a Medtronic Select Secure 3830 pacing lead will be positioned at the His bundle. If selective direct His bundle pacing cannot be achieved then non-selective His bundle pacing will be accepted. AV delay optimisation: will be performed using acute non-invasive blood pressure acquired using the Finometer device (Finapres Medical systems, Netherlands).
Arm/Group | Arm A: Pacing Followed by No-Pacing | Arm B: No-Pacing Followed by Pacing
Number analyzed (Participants) | 83 | 84
% (of time over period)
  M6: number analyzed (Participants) | 74 | 82
  M6 | 90.8 (19.42) | 0 (0)
  M12: number analyzed (Participants) | 70 | 74
  M12 | 1.4 (11.59) | 93.5 (16.48)

7. Secondary Outcome: Changes in Arrythmia Burden (%).
Description: Measured upon completion of run-in (as baseline) and periods 1 & 2 (M6 & M12). Device detected Atrial Fibrillation/Supraventricular Tachycardia (AF/SVT) burden recorded as a percentage of time over the 6-month treatment period.
  Results are descriptive and displayed by treatment and by period.
Time Frame: Baseline, 6 months and 12 months post randomisation.
Population: ITT - Note that results are presented per sequence (e.g, by arm per study period) due to the nature of this particular endpoint.
Measure: Mean (Standard Deviation); unit: % (time under AF/SVT burden)
Arm/Group | Arm A: Pacing Followed by No-Pacing | Arm B: No-Pacing Followed by Pacing
Number analyzed (Participants) | 83 | 84
% (time under AF/SVT burden)
  BL (Randomisation) | 0.1 (0.52) | 0.3 (2.40)
  M6: number analyzed (Participants) | 73 | 80
  M6 | 0.2 (0.62) | 0.1 (0.46)
  M12: number analyzed (Participants) | 70 | 71
  M12 | 0.4 (2.01) | 1.5 (11.87)

8. Secondary Outcome: Changes in Pacing Thresholds (Volts).
Description: Measured upon completion of run-in and periods 1 & 2 (BL, M6 & M12)
  Results are descriptive and displayed by treatment and by period. Please also note that voltage is presented for both RA Lead and LV Lead.
Time Frame: Baseline, 6 months and 12 months post randomisation.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Volts
Arm/Group | Arm A: Pacing Followed by No-Pacing | Arm B: No-Pacing Followed by Pacing
Number analyzed (Participants) | 83 | 84
Volts
  RA Lead - BL: number analyzed (Participants) | 80 | 83
  RA Lead - BL | 0.82 (0.972) | 0.78 (0.510)
  RA Lead - M6: number analyzed (Participants) | 72 | 78
  RA Lead - M6 | 0.82 (1.090) | 0.74 (0.645)
  RA Lead - M12: number analyzed (Participants) | 68 | 71
  RA Lead - M12 | 0.78 (1.034) | 0.79 (0.938)
  LV Lead - BL: number analyzed (Participants) | 82 | 83
  LV Lead - BL | 0.78 (0.438) | 0.84 (0.516)
  LV Lead - M6: number analyzed (Participants) | 74 | 78
  LV Lead - M6 | 0.78 (0.452) | 0.73 (0.265)
  LV Lead - M12: number analyzed (Participants) | 68 | 71
  LV Lead - M12 | 0.78 (0.359) | 0.76 (0.280)

9. Secondary Outcome: Changes in R Wave Amplitude.
Description: Measured from electrocardiogram (ECG).
Time Frame: Baseline, 6 months and 12 months post randomisation.
Population: Null analysis population as r-wave data was unable to be collected
Arm/Group | Arm A: Pacing Followed by No-Pacing | Arm B: No-Pacing Followed by Pacing
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Changes in Lead Impedance (Ohms).
Description: Measured upon completion of run-in and periods 1 & 2 (BL, M6 & M12).
  Results are descriptive and displayed by treatment and by period. Please also note that lead impedance is presented for both RA Lead, HIS-Lead and LV Lead.
Time Frame: Baseline, 6 months and 12 months post randomisation.
Population: - Note that results are presented per sequence (e.g, by arm per study period) due to the nature of this particular endpoint.
Measure: Mean (Standard Deviation); unit: ohms
Arm/Group | Arm A: Pacing Followed by No-Pacing | Arm B: No-Pacing Followed by Pacing
Number analyzed (Participants) | 83 | 84
ohms
  RA Lead Impedance - BL | 460.8 (66.7) | 480.8 (89.24)
  RA Lead Impedance - M6: number analyzed (Participants) | 74 | 81
  RA Lead Impedance - M6 | 475.2 (62.44) | 469.1 (86.48)
  RA Lead Impedance - M12: number analyzed (Participants) | 70 | 72
  RA Lead Impedance - M12 | 452.0 (68.38) | 473.7 (110.6)
  His Lead Impedance - BL: number analyzed (Participants) | 82 | 83
  His Lead Impedance - BL | 377.9 (104.28) | 392.4 (97.94)
  His Lead Impedance - M6: number analyzed (Participants) | 73 | 81
  His Lead Impedance - M6 | 326.3 (84.24) | 326.8 (87.08)
  His Lead Impedance - M12: number analyzed (Participants) | 69 | 72
  His Lead Impedance - M12 | 324.9 (87.08) | 330.6 (82.68)
  LV Lead Impedance - BL: number analyzed (Participants) | 83 | 83
  LV Lead Impedance - BL | 436.5 (90.85) | 464.8 (101.62)
  LV Lead Impedance - M6: number analyzed (Participants) | 74 | 81
  LV Lead Impedance - M6 | 427.8 (87.01) | 439.1 (109.44)
  LVLead Impedance - M12: number analyzed (Participants) | 69 | 72
  LVLead Impedance - M12 | 425.8 (85.06) | 431.2 (9.02)

11. Secondary Outcome: Fluoroscopy Time During Device Insertion.
Description: Measured by time in minutes.
Time Frame: Taken at Device Insertion Visit (2). Baseline measure.
Population: ITT - Note that 2 patients (1 in each arm) have missing data. This outcome measure is only based on the device insertion and does not have a cross-over element.
Measure: Median (Inter-Quartile Range); unit: minutes
Groups:
- Arm A: Pacing Followed by No-Pacing: Device insertion time for those allocated to Arm A
- Arm B: No-Pacing Followed by Pacing: Device insertion time for those allocated to Arm B
Arm/Group | Arm A: Pacing Followed by No-Pacing | Arm B: No-Pacing Followed by Pacing
Number analyzed (Participants) | 82 | 83
minutes | 16.5 [10 to 27] | 16.0 [10 to 26]

12. Secondary Outcome: Changes in Quality of Life Scores. - EQ5D Health State Score
Description: Taken from the Visual Analog Scale (VAS) Score from EQ5D Health State Question in EuroQol, 5-dimension, 5-level (EQ5D5L) questionnaire.
  Score is on a 0-100 scale with 100 representing a better outcome for patients health state.
Time Frame: Baseline, 6 months and 12 months post randomisation.
Population: ITT - Note that some patients were not able to be analysed due to providing no questionnaire data.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Pacing | No-Pacing
Number analyzed (Participants) | 151 | 151
scores on a scale | 66.3 [61.0 to 71.6] | 64.3 [60.4 to 68.3]

ADVERSE EVENTS:
Time Frame: AE Data presented was collected during the treatment phase of the study. 12 months in total.
Description: Please note that due to patient withdrawal prior to period 2 (crossover), the total at-risk population for each arm will be lower than 167.
  Due to withdrawals by period 2, total at risk for Pacing treatment = 160 Due to withdrawals by period 2, total at risk for No-Pacing treatment = 157
  All AEs/SAEs/Mortality events are based on the anticipated treatment being administered during that study period as per randomization arm
Groups:
- Run-in Period (Pre-Randomisation): 2-month run-in period post device implantation. Device switched to no pacing during this period.
- AV Optimised Direct His-bundle (ARM A at Period 1, ARM B at Period 2): Adverse Events & Mortality grouped by treatment received over the 12-month follow-up period. AV optimised direct His-bundle (ARM A at Period 1, ARM B at Period 2).
  Note: Due to withdrawals by period 2, total at risk for Pacing treatment = 160
- No Pacing (ARM A at Period 2, ARM B at Period 1): Adverse Events & Mortality grouped by treatment received over the 12-month follow-up period. No Pacing (ARM A at Period 2, ARM B at Period 1)
  Note: Due to withdrawals by period 2, total at risk for No-Pacing treatment = 157
Arm/Group | Run-in Period (Pre-Randomisation) | AV Optimised Direct His-bundle (ARM A at Period 1, ARM B at Period 2) | No Pacing (ARM A at Period 2, ARM B at Period 1)
All-Cause Mortality (participants affected / at risk) | 0/167 | 6/160 | 4/157
Serious Adverse Events (participants affected / at risk) | 25/167 | 25/160 | 20/157
Other Adverse Events (participants affected / at risk) | 54/167 | 75/160 | 75/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in Period (Pre-Randomisation) (N=167) | AV Optimised Direct His-bundle (ARM A at Period 1, ARM B at Period 2) (N=160) | No Pacing (ARM A at Period 2, ARM B at Period 1) (N=157)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Acute pulmonary oedema and Aortic valve stenosis with insufficiency (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
Atrial arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 3 (3) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Breathlessness (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1) — Exacerbation of heart failure
Cardiac Arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiogenic Shock (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
ICD trigger VF arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Community Acquired Pneumonia (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
Complete Heart Block (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Decompensated / Congestive Cardiac Failure (Cardiac disorders) | 3 (3) | 3 (3) | 8 (8)
Exacerbation of Heart Failure (Cardiac disorders) | 2 (2) | 7 (7) | 2 (2)
Ulcerated legs (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Fluid overload (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
His Lead displacement (Product Issues) | 5 (5) | 1 (1) | 0 (0)
ICD shock (Product Issues) | 2 (2) | 0 (0) | 1 (2)
LRTI (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Haematoma (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Anaphylactic Reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Kidney Disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) — Acute on Chronic Kidney Disease
AKI (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Raised His Lead Threshold (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Subclavian vein thrombosis. (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
VT Episodes (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in Period (Pre-Randomisation) (N=167) | AV Optimised Direct His-bundle (ARM A at Period 1, ARM B at Period 2) (N=160) | No Pacing (ARM A at Period 2, ARM B at Period 1) (N=157)
abnormal blood sugar levels (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Abnormal LFTs (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Accidental morphine overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Acute Kidney Injury (Endocrine disorders) | 0 (0) | 2 (2) | 1 (1)
Ascites (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 6 (6) | 4 (4) | 5 (5)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Baker's cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bilateral leg cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bilateral numbness of arm when lying either side (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Bilateral Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Bloatedness (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Blocked urethral catheter (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac symptoms of palpitations and hypotension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chest Infection (Infections and infestations) | 3 (3) | 9 (12) | 6 (7)
Chest Pain (Cardiac disorders) | 2 (2) | 5 (5) | 4 (4)
Common Colds (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Decompensated Heart Failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic Left Foot Ulcer (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dizziness (General disorders) | 4 (4) | 1 (1) | 2 (2)
Dry persistent cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema Skin condition (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Exacerbation of asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Exacerbation of HF (Cardiac disorders) | 1 (1) | 3 (3) | 5 (5)
Extreme tiredness and fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1)
Fall secondary to dizziness (General disorders) | 2 (2) | 1 (1) | 0 (0)
Feeling of generally unwell (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Fractured foot (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 2 (2)
Haematuria secondary to NOAC (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
HIS lead threshold rise (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Hospital Acquired Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hypergylcaemic Episode (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
Hyperkalaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Idiopathic skin condition (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Impacted ear wax (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Increased breathlessness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 5 (5)
Intermittent cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Laceration to big toe (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Left eye vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Left Kidney Stones (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Mechanical Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
mouth ulcer requiring biopsy (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
New diagnosis of diabetes (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Non cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
nonblanching petechial rashes on both shins (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Non-sustained VT Episodes (Cardiac disorders) | 0 (0) | 6 (6) | 6 (6)
Painful bilateral knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
painful lower extremeties (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Paroxysmal Atrial Fibrillation (Cardiac disorders) | 0 (0) | 4 (4) | 3 (3)
Polyps in colon (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4)
Progressive weight loss (General disorders) | 0 (0) | 1 (1) | 0 (0)
Raised His Lead Threshold (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Raised INR (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Received external electrical shock at work (works as an electrician) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
recurrence of atrial arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Recurrence of atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Shortness of breath, Productive cough and wheeze due to lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
skin cancer growth L) hand (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Sprained wrist due to fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Suspected lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sustained VT treated with ATP (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
swollen abdomen (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
swollen bilateral legs (knee to ankle) (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Swollen feet (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Swollen left arm secondary to blood clot (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thyroid Deficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 3 (3) | 2 (2)
Ventricular Tachycardia Episodes (Cardiac disorders) | 6 (6) | 5 (5) | 2 (2)
Viral Illness of unknown origin (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Weight loss and dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Worsening chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Worsening renal function (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
worsening shortness of breath and activity tolerance (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Shortness of breath secondary to bilateral pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
LRTI (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Anterior L1 Compression Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Barrett's Oesophagus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bilateral swollen and painful legs (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Broken rib (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Cataracts operation on left eye (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Coronary Sinus lead displaced (Product Issues) | 0 (0) | 0 (0) | 1 (1)
decreased activity tolerance and increased paroxysmal nocturnal dyspnea (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Degenerated rotator cuff and tendinopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Dislocated R shoulder due to mechanical fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Excessive intestinal gas -belching or flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fainting spells (General disorders) | 0 (0) | 0 (0) | 2 (2)
Fall. Walking sticks slipped off. (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1)
Fracture in left elbow due to a fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Heartburn (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Heavily trabeculated bladder with debris in urine noted during flexible cystoscopy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Increased urinary frequency secondary to enlarged prostate (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
insertion of indwelling catheter (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Intermittent high impedance on His Lead with increase in His pacing threshold (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Late His Lead threshold rise (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Left leg cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Left lower leg blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
left ventricular thrombus (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Lesion in caecum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Marked deterioration of kidney function (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Mild Infective Exacerbation of Bronchiectasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
MRSA positive nose and groin (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Non-tender pain free lump increasing in size (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Recurrent Falls secondary to hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Progressive worsening of breathlessness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Reduced mobility (General disorders) | 0 (0) | 0 (0) | 1 (1)
Right leg cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Shoulder joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Slight palpitations, Chest discomfort. (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ST elevation on ECG post MVO2 (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Swollen right leg ?secondary to blood clot (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
TIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tingling sensation in both feet (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
worsening shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peptic Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Endoscopy (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Blood and lymphatic system disorders) | 5 (5) | 0 (0) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
URTI (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vasovagal episode (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Ventricular Ectopy burden (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Injury due to Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
High atrial lead threshold (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hives (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension and dizziness (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Mixed anaerobes in catheter swab (Investigations) | 1 (1) | 0 (0) | 0 (0)
Adverse chest findings following x-ray (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nitrites in Urine (Investigations) | 1 (1) | 0 (0) | 0 (0)
Pseudomonas in urine (Investigations) | 1 (1) | 0 (0) | 0 (0)
Seroma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
serous fluid found in old generator box site (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Pleural Effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular Ectopy burden (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Low QRS Duration (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pain and limited mobility in the arm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT02671903/Prot_001.pdf
  • Statistical Analysis Plan (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT02671903/SAP_000.pdf